CLINICAL TRIAL: NCT00462592
Title: A Randomised Double Blind, Placebo Controlled 4-way Cross Over Study Comparing Montelukast, Inhaled Budesonide and Their Combination on Exercise-induced Bronchoconstriction
Brief Title: Comparison of Combination Therapy: Montelukast and Inhaled Steroid on Exercise Induced Bronchoconstriction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Paul O'Byrne, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: monbud8035
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Asthma
Keywords: exercise-induced bronchoconstriction (EIB); airway inflammation
MeSH Terms: conditions — Asthma | interventions — Budesonide; montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): montelukast - montelukast 5 mg ( < 15 years) or 10 mg (and matching placebo)will be taken 1 tab in the evening
  Interventions: Drug: montelukast; Other: placebo
- 2 (Active Comparator): budesonide - inhaled budesonide turbuhaler 200ug (& matching placebo) taken 1 puff morning & 1 puff evening.
  Interventions: Drug: budesonide; Other: placebo
- 3 (Placebo Comparator): placebo
  Interventions: Other: placebo
- 4 (Active Comparator): montelukast budesonide combination - montelukast 5mg ( < 15 years) or 10 mg (& matching placebo)will be taken 1 tab in the evening together with inhaled budesonide turbuhaler 200 ug (& matching placebo) taken 1 puff morning & 1 puff evening.
  Interventions: Drug: budesonide; Drug: montelukast; Other: placebo

INTERVENTIONS:
Drug: budesonide — inhaled budesonide turbuhaler 200ug taken 1 puff morning & 1 puff evening.
  Other Names: budesonide (Pulmicort)
  Arms: 2; 4
Drug: montelukast — montelukast 5 mg ( < 15 years) or 10 mg (and matching placebo)will be taken 1 tab in the evening
  Other Names: montelukast (Singulair)
  Arms: 1; 4
Other: placebo — placebo

SUMMARY:
The purpose of this study is to compare the effects of 2 weeks therapy of montelukast, budesonide, their combination on exercise induced bronchoconstriction (EIB) and airway inflammation in children and young adults, not on regular controller therapy.

Inhaled corticosteroids (ICS) are potent anti-inflammatory agents, which are effective in controlling and improving all aspects of asthma including the attenuation of EIB. However, the effect of ICS monotherapy on EIB is comparable if not inferior to the effect of CysLTs modifiers alone. This may be due to the lack of effect of ICS on the CysLT pathway. As a consequence, the investigators hypothesize that the combination of ICS and CysLT modifiers will offer a greater protection against EIB than either therapy alone. The different classes of drugs may act on complementary pathways believed to be important in the pathophysiology of EIB.

DETAILED DESCRIPTION:
The study will be a 2 centre randomised, double blind, placebo controlled 4-way cross over study comparing montelukast, budesonide and their combination on exercise-induced bronchoconstriction (EIB). Subjects with stable mild to moderate asthma, between the ages of 8-35 years, not on controller asthma therapy will be screened. A maxFEV1% ≥15% following a standardized dry air exercise challenge at screening (SC) and following a 1 week run-in (V-1) is required to qualify. Once qualified, subjects will return the following day (V0) for a skin prick test and a methacholine inhalation test before being randomised to 1 of 4 treatment sequences. Each treatment will be given for a total of 14 days with a 4 weeks washout. During each period, subjects will attend the laboratory on 2 occasions, at the beginning and end of each period. Baseline spirometry; eNO; EBC will be performed, followed by an exercise challenge with serial FEV1 and eNO measurements up to 30 minutes post exercise and post-exercise EBC and sputum induction at each evaluation visit. There will be a total of 10 visits and the duration of study will be approximately 148 days (21 weeks). All visits will be scheduled within 2 hours of the post-run visit (V1) and at least 8 hours after the last dose of trial medications.

Investigational Product, Dose and Administration:

Montelukast 5mg (<15 years) or 10mg (and matching placebo) will be taken 1 tablet in the evening together with inhaled budesonide turbuhalers 200ug (and matching placebo) taken 1 puff in the morning and 1 puff in the evening.

Efficacy on EIB:

The changes between pre and post treatment exercise-induced maxFEV1% and area under the curve (AUC0-30) will be compared between the 4 periods. MaxFEV1% will be calculated as pre-exercise FEV1 minus post exercise lowest FEV1 divided by pre-exercise FEV1 multiplied by 100; AUC will be calculated using the trapezoidal rule. The protection provided by the active treatments will be defined as the pre-treatment maxFEV1% minus post-treatment maxFEV1% divided by pre-treatment maxFEV1% x 100. The proportions of subjects attaining ≥50% protection will be compared between the 4 arms.

Efficacy on eNO and inflammatory parameters measured in sputum and EBC Changes in % and absolute counts of sputum differential cells, eNO and inflammatory mediators (in EBC/ sputum) at baseline and in response to exercise will be compared between the 4 arms.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 8-35 years with stable mild-to-moderate asthma (ATS criteria) not on regular controller therapy
* Prebronchodilator FEV1 predicted ≥ 70%
* No other medical co-morbidity
* Demonstrate maxFEV1% ≥15% on exercise challenge at screening and 1 week post run-in.

Exclusion Criteria:

* Asthma exacerbations or respiratory infection within 4 weeks of screening
* Recent use of inhaled or systemic steroids
* Immunosuppressives
* Antihistamines, NSAIDs and investigational drugs within 30 days
* Unable to reliably perform spirometry and exercise challenge
* Current or ex-smokers ≥ 10 pack-years and less than 1 month abstinence
* Contra-indications to inhaled steroids or montelukast use.

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The magnitude of protection and the number of subjects with ≥50% protection (considered to be clinically relevant) following treatment | Before and after 2 weeks of treatment in each 4 arm

SECONDARY OUTCOMES:
Change in sputum cell counts and fluid phase inflammatory mediators | Before and after 2 weeks of treatment in each 4 arm
Change in baseline exhaled nitric oxide (eNO) and response to exercise challenge | Before and after 2 weeks of treatment in each 4 arm
Change in EBC (exhaled breath condensate) inflammatory mediators from baseline | Before and after 2 weeks of treatment in each 4 arm
The change in exercise induced maximal percent fall in FEV1 (maxFEV1%) and area under the curve (AUC0-30) relative to pre-exercise FEV1 up to 30 minutes following exercise challenge | Before and after 2 weeks of treatment in each 4 arm

CONTACTS AND LOCATIONS:
Overall Officials: Paul O'Byrne, MD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Hamilton Health Sciences-McMaster University, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario